CLINICAL TRIAL: NCT07157592
Title: The Effect of Ventrogluteal Intramuscular Injection Technique on Pain and Physiological Parameters in Children: A Quasi-Experimental Study
Brief Title: Effect of Ventrogluteal Intramuscular Injection Technique on Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Banu Terzi, Banu Terzi, PhD, RN, Associate Professor, Akdeniz University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023/06
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: IM Injection; Ventrogluteal Site; Children; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ventrogluteal IM injection protocol (Experimental)
  Interventions: Other: Ventrogluteal IM Injection tecnique

INTERVENTIONS:
Other: Ventrogluteal IM Injection tecnique — Ventrogluteal IM injection technique:
  During IM injection into the ventrogluteal region:
  * The entrance angle of the needle is 90º.
  * The 25-gauge (1-inch) syringe is held with the active hand as if holding a pen, and no hand change is made during the injection.
  * The needle is rapidly inserted into the skin and withdrawn at the same angle 5 seconds after the injection.
  * The drug is injected for 5 seconds/mL without blood aspiration during injection.
  * Light pressure is applied to the area after injection, with no massage performed.
  To evaluate the appropriateness of the application ventrogluteal IM injection technique, the opinions were obtained of five experts in nursing principles and child health and disease nursing.

SUMMARY:
Intramuscular injection is one of the most frequently practiced basic nursing skills in emergency units. However, serious complications may develop when this skill is not applied with the correct technique.

The aim of the study is to investigate the effect of ventrogluteal intramuscular injection technique on pain and physiological parameters in children.

The quasi-experimental study was conducted with 90 children aged 6-12 years. The data were obtained from two groups: the control group, in which routine care was applied during intramuscular injection, and the intervention group, in which the ventrogluteal intramuscular injection technique was applied. The pain and physiological parameters of children in both groups before and after the intervention were compared.

The mean pulse rate was lower in the intervention group compared to the control group after the procedure (p<0.05). When the mean pain scores after the procedure were analyzed, the scores in the intervention group were lower than in the control group (p<0.05). The use of ventrogluteal intramuscular injection technique during in children was effective in reducing pain levels and decreasing pulse rate. These findings support incorporating this technique into routine nursing practice to enhance comfort and safety during intramuscular injections in children.

ELIGIBILITY:
Inclusion Criteria:

* Being 6-12 years old.
* Being willing to participate in the research.
* Not having a chronic disease or mental or neurological disability.
* Being able to communicate verbally.

Exclusion Criteria:

* Taking any analgesic medication within 6 hours before the application to the emergency department.
* Having a life-threatening disease (e.g., sepsis, shock, respiratory or cardiogenic arrest).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Wong-Baker Scale (Pain Face Rating Scale) | Before and 5 minutes after the procedure
  Faces represent increasing pain intensity from 0 to 5 from left to right. The leftmost face has a smiling expression indicating a pain-free state, whereas the face at the right end has a crying expression corresponding to the most severe pain. Below each face is a short description of the pain intensity: 0-no pain, 1-mild pain, 2-slightly more pain, 3-even more pain, 4-considerably more pain, and 5-most severe pain
SpO2 and pulse rate | Before and 5 minutes after the procedure
  A calibrated pulse oximeter (Nellcor OxiMax N-65) was used to determine the oxygen saturation (SpO2) and pulse rate of the children before and after vaccine injection. The pulse oximeter shows the SpO2 and pulse rate on an LCD screen. It works with four AA batteries. The SpO2 and pulse rate were obtained by attaching the probe of the pulse oximeter to the thumb of the children.
Blood pressure | Before and 5 minutes after the procedure
  A calibrated digital sphygmomanometer (Omron M3 Comfort) was used to determine the blood pressure of the children before and after IM injection. The sphygmomanometer shows systolic and diastolic blood pressure values on an LCD screen. A baby cuff was attached to the sphygmomanometer, and the systolic and diastolic blood pressure values were determined by attaching the cuff to the right arm of the children.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No